CLINICAL TRIAL: NCT00661557
Title: Immunogenicity & Safety Study of GSK Biologicals' Meningococcal Vaccine GSK134612 Administered in Healthy Subjects Either Previously Primed With Mencevax™ ACWY or naïve to Meningococcal Vaccination.
Brief Title: Comparison of GSK134612 in Subjects Previously Vaccinated Against Meningococcal Disease Versus Non-vaccinated Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107408
Record Dates: First submitted 2008-04-14; First posted 2008-04-18 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-06

CONDITIONS: Infections, Meningococcal
Keywords: Booster vaccination; Meningococcal vaccine; Meningococcal disease; Safety; immunogenicity
MeSH Terms: conditions — Meningococcal Infections

ARMS (2):
- Mencevax Primed Group (Experimental): Subjects who were previously vaccinated with meningococcal vaccine Mencevax ACWY in study NCT00227422 received in the current study a single dose of meningococcal conjugate vaccine Nimenrix, administered intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Meningococcal vaccine GSK134612 (Nimenrix)
- Mencevax Naive Group (Active Comparator): Subjects who did not receive (or had not received in the preceding 10 years) any meningococcal vaccination received in the current study a single dose of meningococcal conjugate vaccine Nimenrix, administered intramuscularly in the deltoid muscle of the non-dominant arm.
  Interventions: Biological: Meningococcal vaccine GSK134612 (Nimenrix)

INTERVENTIONS:
Biological: Meningococcal vaccine GSK134612 (Nimenrix) — one dose, as intramuscular injection

SUMMARY:
In this study, subjects who were vaccinated with a meningococcal polysaccharide vaccine in a previous study (whose objectives & outcome measures are presented in a separate protocol posting with NCT number = 00227422) will be vaccinated with a new vaccine using conjugation technology.

These subjects will be compared to subjects vaccinated with the new vaccine, but who were not previously vaccinated with a meningococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
GSK Biologicals has developed a meningococcal conjugate vaccine (GSK134612). This candidate vaccine has been shown to be well tolerated and immunogenic in toddlers, children aged 3-5 years, and adolescents/young adults. Repeated vaccinations with unconjugated meningococcal polysaccharide vaccine has shown to induce hyporesponsiveness to re-vaccination, this for serogroup C, and a recent publication suggest the same may be true for other serogroups.

This study will evaluate GSK Biologicals' candidate vaccine's ability to induce satisfactory immune response for the serogroups it contains across subjects 4.5 through 34 years of age who previously received a tetravalent meningococcal polysaccharide vaccine when aged 2-30 years. A non-randomised age-strata matched group of subjects, who have not previously received (or not received within the preceding 10 years) any meningococcal vaccine, will also be administered the GSK134612 vaccine for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects who the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* For the MPS group, a male or female between, and including, 4.5 and 34 years of age at the time of the study vaccination, who has been vaccinated in GSK Biologicals' study 102394.
* For the noMPS group, a male or female between, and including, 4.5 and 34 years of age at the time of the study vaccination.
* Written informed consent obtained from the subject/ from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her knowledge.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding administration of the study vaccine, or planned use during the complete study period (active phase and extended safety follow-up).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the study vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of administration of the study vaccine and up to 30 days after the study vaccine.
* Concurrently participating in another clinical study, at any time during the study period (active phase and extended safety follow-up), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* For the MPS Group, vaccination against meningococcal disease after completion of study 102394
* For the noMPS group, previous vaccination, or vaccination within the last 10 years, against meningococcal disease (of any serogroup).
* Previous vaccination against tetanus within 30 days.
* History of meningococcal disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, based on medical history and physical.
* A family history of congenital or hereditary immunodeficiency, unless the child has previously been documented, through laboratory testing, to have normal immune function.
* History of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* Know hypersensitivity to any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of seizures (this criterion does not apply to subjects who have had a single, uncomplicated febrile convulsion in the past) or progressive neurological disease.
* Acute disease at the time of enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the active stage of the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.

Ages: 4 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 271 (Actual)
Dates: Start 2008-05-19 (Actual); Primary Completion 2008-12-19 (Actual); Study Completion 2008-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dbaibo G, Van der Wielen M, Reda M, Medlej F, Tabet C, Boutriau D, Sumbul A, Anis S, Miller JM. The tetravalent meningococcal serogroups A, C, W-135, and Y tetanus toxoid conjugate vaccine is immunogenic with a clinically acceptable safety profile in subjects previously vaccinated with a tetravalent polysaccharide vaccine. Int J Infect Dis. 2012 Aug;16(8):e608-15. doi: 10.1016/j.ijid.2012.04.006. Epub 2012 Jun 14. PMID 22704725
- [Background] Dbaibo G et al. One dose of the meningococcal tetravalent tetanus toxoid conjugated vaccine (MenACWY-TT) is immunogenic with an acceptable safety profile in unvaccinated subjects and those previously vaccinated with a MenACWY polysaccharide vaccine. Abstract presented at the 3rd Northern European Conference on Travel Medicine (NECTM). Hamburg, Germany, 26-29 May 2010.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 107408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Started | 192 | 79
Completed | 183 | 79
Not Completed | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mencevax Primed Group | Mencevax Naive Group | Total
Number analyzed (Participants) | 192 | 79 | 271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.1 (6.79) | 14.2 (7.23) | 14.13 (6.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 41 | 132
  Male | 101 | 38 | 139
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Arabic/North African heritage | 192 | 77 | 269
  White - Caucasian/European heritage | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Meningococcal Serum Bactericidal Antibodies/Assay (rSBA) Titers
Description: For each antibody assessed (serogroups A, C, W, and Y) at the corresponding time point, titers were expressed as geometric mean titers (GMTs) and tabulated with 95% confidence intervals (CIs).
Time Frame: One month post-vaccination (Month 1)
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variable measures at the defined timepoint were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 169 | 75
Titers
  rSBA-MenA: number analyzed (Participants) | 146 | 69
  rSBA-MenA | 6868.8 [6044.9 to 7805.0] | 13014.9 [10722.2 to 15798.0]
  rSBA-MenC | 1945.8 [1583.3 to 2391.1] | 5494.6 [4266.3 to 7076.5]
  rSBA-MenW-135 | 4635.7 [3942.5 to 5450.7] | 9078.0 [7087.7 to 11627.1]
  rSBA-MenY: number analyzed (Participants) | 167 | 75
  rSBA-MenY | 7799.9 [6682.8 to 9103.6] | 13895.5 [11186.2 to 17260.9]

2. Secondary Outcome: Meningococcal rSBA Titers
Description: as for outcome 1
Time Frame: Prior to vaccination (Day 0)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 167 | 74
Titers
  rSBA-MenA: number analyzed (Participants) | 160 | 71
  rSBA-MenA | 1770.1 [1569.0 to 1996.9] | 1103.8 [863.2 to 1411.5]
  rSBA-MenC: number analyzed (Participants) | 165 | 70
  rSBA-MenC | 116.6 [80.2 to 169.4] | 30.1 [17.4 to 52.0]
  rSBA-MenW-135: number analyzed (Participants) | 165 | 74
  rSBA-MenW-135 | 154.0 [114.0 to 208.1] | 36.9 [22.7 to 59.9]
  rSBA-MenY | 555.2 [434.8 to 708.9] | 170.1 [106.1 to 272.9]

3. Secondary Outcome: Anti-meningococcal Polysaccharide (PS) Antibody Concentrations
Description: For each antibody assessed (serogroups A, C, W, and Y) at the corresponding time point, polysaccharide antibody concentrations were expressed as geometric mean concentrations (GMCs) in micrograms per milliliter (µg/mL) and tabulated with 95% confidence intervals (CIs).
Time Frame: Prior to (Day 0) and one month post-vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 86 | 38
µg/mL
  Anti-PSA, Day 0: number analyzed (Participants) | 82 | 38
  Anti-PSA, Day 0 | 9.38 [6.37 to 13.81] | 0.41 [0.24 to 0.70]
  Anti-PSA, Month 1: number analyzed (Participants) | 82 | 38
  Anti-PSA, Month 1 | 79.15 [57.61 to 108.73] | 47.45 [30.48 to 73.85]
  Anti-PSC, Day 0: number analyzed (Participants) | 82 | 38
  Anti-PSC, Day 0 | 6.46 [4.49 to 9.30] | 0.31 [0.20 to 0.47]
  Anti-PSC, Month 1: number analyzed (Participants) | 82 | 38
  Anti-PSC, Month 1 | 31.19 [25.34 to 38.39] | 18.81 [12.92 to 27.38]
  Anti-PSW-135, Day 0: number analyzed (Participants) | 76 | 35
  Anti-PSW-135, Day 0 | 3.40 [2.20 to 5.26] | 0.20 [0.14 to 0.29]
  Anti-PSW-135, Month 1: number analyzed (Participants) | 85 | 37
  Anti-PSW-135, Month 1 | 25.10 [19.49 to 32.33] | 14.67 [9.25 to 23.28]
  Anti-PSY, Day 0: number analyzed (Participants) | 85 | 36
  Anti-PSY, Day 0 | 4.05 [2.83 to 5.81] | 0.21 [0.15 to 0.29]
  Anti-PSY, Month 1: number analyzed (Participants) | 86 | 37
  Anti-PSY, Month 1 | 29.98 [23.48 to 38.28] | 17.58 [11.89 to 25.99]

4. Secondary Outcome: Anti-tetanus Toxoid Antibody Concentrations
Description: Antibody concentrations were tabulated as geometric mean concentrations (GMCs) in International Units per milliliter (IU/mL), with 95% confidence intervals (CIs).
Time Frame: Prior to (Day 0) and one month post-vaccination (Month 1)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 169 | 75
IU/mL
  Pre-vaccination | 0.718 [0.561 to 0.919] | 1.515 [1.032 to 2.223]
  Post-vaccination | 17.678 [14.494 to 21.562] | 41.600 [31.587 to 54.787]

5. Secondary Outcome: Number of Subjects With a Vaccine Response to Meningococcal Antigens A, C, W and Y
Description: Vaccine response defined as:
  For initially seronegative subjects: post-vaccination antibody titer ≥1:32 For initially seropositive subjects: post-vaccination antibody titer ≥4-fold the pre-vaccination antibody titer
Time Frame: One month post-vaccination (Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 167 | 74
Participants
  rSBA-MenA: number analyzed (Participants) | 141 | 65
  rSBA-MenA | 58 | 50
  rSBA-MenC: number analyzed (Participants) | 165 | 70
  rSBA-MenC | 110 | 68
  rSBA-MenW-135: number analyzed (Participants) | 165 | 74
  rSBA-MenW-135 | 137 | 72
  rSBA-MenY | 125 | 71

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 4-day (Day 0 to Day 3) period after vaccination
Population: This analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects. Only subjects who completed their symptom sheets are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 165 | 77
Participants
  Any Pain | 84 | 27
  Grade 3 Pain | 8 | 0
  Any Redness | 35 | 17
  Grade 3 Redness | 3 | 1
  Any Swelling | 40 | 20
  Grade 3 Swelling | 9 | 2

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], headache, myalgia, shivering and sweating. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Day 0 to Day 3) period after vaccination
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 165 | 77
Participants
  Any Fatigue | 59 | 15
  Grade 3 Fatigue | 9 | 2
  Related Fatigue | 54 | 9
  Any Fever (oral temperature) | 33 | 15
  Grade 3 Fever (oral temperature) | 2 | 0
  Related Fever (oral temperature) | 31 | 6
  Any Gastrointestinal Symptoms | 26 | 10
  Grade 3 Gastrointestinal Symptoms | 4 | 0
  Related Gastrointestinal Symptoms | 24 | 6
  Any Headache | 52 | 17
  Grade 3 Headache | 5 | 0
  Related Headache | 45 | 9

8. Secondary Outcome: Number of Subjects With Unsolicited Symptoms
Description: An unsolicited symptom covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: Up to one month post-vaccination (Month 1)
Population: This analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 192 | 79
Participants | 19 | 11

9. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Day 0 to study month 6
Population: This analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 192 | 79
Participants | 1 | 0

10. Secondary Outcome: Number of Subjects With Any Specific Adverse Events
Description: Specific adverse events comprised rash, new onset of chronic illnesses (NOCIs), conditions prompting emergency room (ER) visits and/or any event related to lack of vaccine efficacy (i.e. documented meningococcal disease).
  Events related to lack of vaccine efficacy (i.e. meningococcal disease) were recorded, but because such events were life threatening and were thus reported as SAEs, these events were not analyzed or reported here separately.
Time Frame: Day 0 to study month 6
Population: This analysis was based on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
Number analyzed (Participants) | 192 | 79
Participants
  Subjects with any rash | 0 | 0
  Subjects with any NOCI(s) | 0 | 2
  Subjects with any ER visit(s) | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms: Day 0 to Day 3 post-vaccination; Unsolicited symptoms: Day 0-Day 30 post-vaccination. Serious adverse events: Day 0 up to study end at Month 6.
Arm/Group | Mencevax Primed Group | Mencevax Naive Group
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/79
Serious Adverse Events (participants affected / at risk) | 1/192 | 0/79
Other Adverse Events (participants affected / at risk) | 111/192 | 42/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mencevax Primed Group (N=192) | Mencevax Naive Group (N=79)
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mencevax Primed Group (N=192) | Mencevax Naive Group (N=79)
Erythema (Skin and subcutaneous tissue disorders) | 35 (35) | 17 (17)
Fatigue (General disorders) | 59 (59) | 15 (15)
Gastrointestinal disorder (Gastrointestinal disorders) | 26 (26) | 10 (10)
Headache (Nervous system disorders) | 53 (53) | 17 (17)
Pain (General disorders) | 84 (85) | 27 (27)
Pyrexia (General disorders) | 34 (34) | 15 (15)
Swelling (General disorders) | 40 (40) | 20 (20)
Tonsillitis (Infections and infestations) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.